CLINICAL TRIAL: NCT00000605
Title: Estrogen and Graft Atherosclerosis Research Trial (EAGER)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 109; 5U01HL050840 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-04

CONDITIONS: Cardiovascular Diseases; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Myocardial Ischemia; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Hormone Replacement Therapy; Estrogens; Medroxyprogesterone

INTERVENTIONS:
Drug: hormone replacement therapy
Drug: estrogens
Drug: medroxyprogesterone

SUMMARY:
To determine if postmenopausal hormone replacement therapy in women following coronary bypass surgery would reduce the occurrence of graft occlusion and delay the development of graft atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary atherosclerosis is a major cause of death in women in the United States. Although coronary artery bypass surgery decreases symptomatic and clinical evidence of ischemia, it does not alter the underlying process. Patients may present several years later with recurrent symptoms that may be a result of occlusion of saphenous vein grafts, development of atherosclerotic disease in vein grafts, or progression of underlying disease. Any intervention that can reduce the rate of progression of coronary atherosclerosis following bypass surgery would provide significant benefit for women following bypass surgery and possibly for other women with atherosclerotic disease. Observational studies suggest that postmenopausal estrogen replacement therapy is associated with a reduction in cardiac morbidity.

DESIGN NARRATIVE:

The study was a randomized, double-blind, controlled trial. Subjects were randomized to conjugated estrogen with daily medroxyprogesterone or placebo within two weeks of bypass surgery. Graft occlusion and development of vein graft atherosclerosis were measured by comparing quantitative coronary angiographic and vascular ultrasonic assessment of disease severity and extent performed at six months and three and a half years after randomization. The primary outcome variables included the occurrence of graft occlusion at six months and the change in severity and extent of atherosclerosis in the saphenous vein grafts over three years. The trial determined the influence of hormone replacement therapy on the primary outcome variables.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Postmenopausal women who had undergone coronary artery bypass graft.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08; Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Ouyang — Johns Hopkins University